CLINICAL TRIAL: NCT04625322
Title: INSPIRE: Interventions for Screening and Treatment of Psychiatric Inpatients With HCV Resulting in Elimination
Brief Title: HCV Treatment Initiation During Acute Psychiatric Admission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5188
Record Dates: First submitted 2020-09-29; First posted 2020-11-12 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Psychiatric; Hospital; Treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Models of Care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Referral to outpatient specialty for HCV care (No Intervention): Acute psychiatric patients who test HCV RNA positive by OraQuick HCV Antibody Test will be referred for outpatient specialty follow-up at the Toronto Centre for Liver Disease (TCLD) where they will be assessed and offered treatment as per standard of care. TCLD referrals are triaged by clinicians unaware of the trial and prioritized based on urgency of treatment. Patients who do not attend the initial visit will be rescheduled. After 3 'no-show' visits, the person will not be scheduled again at TCLD and will be deemed a 'treatment failure' for the trial with subsequent HCV follow-up at the discretion of the CAMH provider, consistent with current practice.
- Receive HCV care during inpatient admission by a hospitalist (Experimental): CAMH hospitalists covering the inpatient units will undergo a training designed for non-specialist providers, used in the ASCEND trial, which has already occurred. An algorithm-based work-up which has been used for non-specialist treaters in ECHO Liver, a Ministry-of-Health supported tele-mentoring program, will then be completed for all who test HCV RNA positive. Labs will be drawn by the hospital phlebotomist following a positive HCV RNA result from the Gene Xpert Viral Load Assay. At this time, a sample will also be obtained to send to for conventional HCV RNA quantification and genotyping.
  Interventions: Other: HCV care provided by hospitalist during acute psychiatric admission

INTERVENTIONS:
Other: HCV care provided by hospitalist during acute psychiatric admission — HCV diagnosis and treatment will be conducted by a hospitalist during an acute psychiatric admission at CAMH
  Arms: Receive HCV care during inpatient admission by a hospitalist

SUMMARY:
Hepatitis C virus (HCV) disproportionally affects certain populations, including those facing substance use and mental health challenges. In the past, many individuals with mental illness were not treated due to the psychiatric side-effects of interferon. However, the development of highly effective, direct-acting antivirals (DAA) has revolutionized HCV treatment such that cure rates are >95% with 8-12 weeks of simple, safe, and well-tolerated therapy.

A recent systematic review reported that across 13 North American studies, HCV prevalence among people admitted to psychiatric hospitals was a staggering 17.4% (13.2-22.6%). Despite these concerning figures, mental health facilities have not been a focus of HCV elimination efforts to date. The Centre for Addiction and Mental Health (CAMH) in Toronto is the largest mental health facility in Canada, with a psychiatric emergency department seeing ~35 patients per day with many admitted to the acute psychiatric units for safety and stabilization. Currently, psychiatric patients screened for HCV at CAMH have a 75% 'no show' rate at the Toronto Centre for Liver Disease (TCLD), which is located less than 5km away, suggesting that referral upon discharge is ineffective.

This study will be the first trial to evaluate whether it would be feasible and beneficial to initiate treatment during an acute psychiatric admission rather than referring to specialty upon discharge. The combination of broad HCV screening with rapid linkage to treatment has led to successful elimination of HCV within defined populations, so-called micro-elimination. The investigators hypothesize that HCV treatment can be effectively delivered by providers in psychiatric care facilities, which will improve treatment uptake over traditional referral models.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HCV infection, positive HCV RNA
2. Aged 18 to 80
3. Willingness and capacity to provide informed consent, or consent is provided by a substitute decision maker

Exclusion Criteria:

1. Presence of or history of decompensated cirrhosis (evidence of decompensation with history of either ascites, variceal hemorrhage, or hepatic encephalopathy)
2. Platelets < 75,000/mm3, total albumin <35 g/L, total bilirubin >34 μmol/L, INR >1.5
3. History of current or past hepatocellular carcinoma.
4. HBV (HBsAg +ve) co-infection or untreated HIV co-infection
5. Prior HCV antiviral therapy with DAA with or without peginterferon/ribavirin
6. Chronic liver disease other than mild nonalcoholic or alcoholic fatty liver disease from a cause other than HCV
7. Pregnancy/breastfeeding/inability to use contraception
8. Use of concomitant contraindicated medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
SVR12 by intention to treat (ITT) in each arm | 24 months
  To determine whether screening for HCV using rapid diagnostics during an acute psychiatric admission with inpatient initiation of HCV treatment is superior to standard post-discharge referral and treatment by intention to treat (ITT).

SECONDARY OUTCOMES:
SVR12 by modified intention to treat (mITT) in each arm | 24 months
  To determine whether screening for HCV using rapid diagnostics during an acute psychiatric admission with inpatient initiation of HCV treatment is superior to standard post-discharge referral and treatment by modified intention to treat (mITT).
HCV relapse rate | 24 months
  To compare the HCV viral relapse rate in both arms (re-appearance of HCV RNA in those undetectable at end of treatment; relapse distinguished from reinfection by sequencing of the recurrent HCV RNA and comparing to baseline).
HCV seroprevalence rates | 12 months
  To determine HCV seroprevalence rates among acute vs addictions patients admitted to CAMH.
HCV RNA positivity rates | 12 months
  To determine HCV RNA positivity rates among acute vs addictions patients admitted to CAMH.
CAMH staff acceptability of POC antibody and RNA testing | 12 months
  CAMH staff involved in the trial will be asked to particiapte in an acceptibility survey regarding rapid POC antibody and RNA testing on the acute units.
Concordance of POC HCV RNA with HCV RNA by phlebotomy | 12 months
  To determine concordance of POC HCV RNA (GeneXpert) with HCV RNA by phlebotomy (Abbott RealTime).
Minimum and mean times from diagnosis to treatment initiation | 24 months
  Evaluate the mean and minimum times to treatment initiation in both arms, and compare.
Adherence with out-patient follow-up visits | 24 months.
  Evaluate and compare out-patient follow-up visit adherence in both arms.
Adherence to HCV treatment, by HCV regimen | 24 months.
  Evaluate and compare both arms for medication adherence (patient self-report and pill count), and variance by medication regimen.
Adverse events while on HCV treatment | 18 months.
  To determine and compare adverse events in both arms while patients are on treatment.
HCV Reinfection | 24 months.
  Reinfection rates by the end of the defined as HCV RNA detectability after prior SVR with demonstration of distinct viral sequence from baseline sample to distinguish

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No